CLINICAL TRIAL: NCT00004496
Title: Phase I Study of Alpha-Melanocyte Stimulating Hormone in Patients With Acute Renal Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Masking: Double | Purpose: Treatment
Other Study IDs: 199/14286; UTSMC-FDR001552; UTSMC-129447100
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-08

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Acute Kidney Injury; Rare Diseases; Urogenital Diseases | interventions — Adrenocorticotropic Hormone

INTERVENTIONS:
Drug: alpha-melanocyte stimulating hormone

SUMMARY:
OBJECTIVES: I. Determine the maximum tolerated dose and safety of alpha-melanocyte stimulating hormone (alpha-MSH) in patients with acute renal failure.

II. Determine the safety and pharmacokinetics of alpha-MSH in patients at high risk of acute renal failure after renal transplantation.

III. Determine the safety and pharmacokinetics of alpha-MSH in patients with established ischemic acute renal failure.

IV. Determine the effect of alpha-MSH on interleukin-10 pharmacokinetics.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a dose escalation, double blind, placebo controlled, multicenter study.

Group 1: Patients are infused with alpha-melanocyte stimulating hormone (alpha-MSH) or placebo over 5 minutes. A cohort of 5 patients is infused at each dose level of alpha-MSH until the minimum effective dose (MED) and the maximum tolerated dose (MTD) are determined.

Group 2: Patients receive a single dose of the MED of alpha-MSH IV over 5 minutes at the time anastomoses are complete. Other patients receive alpha-MSH at the MTD. Cohorts of 5 patients each are treated at the MED and the MTD.

Group 3: Patients receive alpha-MSH as in group 2. Additional dose levels are also tested.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Group 1: Patients on chronic hemodialysis

Group 2: Patients at high risk of developing acute renal failure (ARF) after cadaveric renal transplantation Received high risk allograft Cadaveric kidneys with greater than 24 hours of cold ischemia time Donor had rising creatinine before organ procurement Donor over 60 years

Group 3: Patients with ischemic ARF due to hypotension, surgery, or trauma ARF severity index 20-60% Creatinine clearance 12-14 mL/min Rising creatinine of at least 0.5 mg/dL per day for 2 days without evidence of recovery despite standard supportive care No drug or contrast induced renal failure No oliguric renal failure (creatinine clearance 3-4 mL/min) No prior chronic renal failure Baseline creatinine greater than 2.5 mg/dL (males) or 2.0 mg/dL (females) No ARF due to bacterial or fungal sepsis, nephrotoxins, acute tubulointerstitial nephritis, cyclosporine toxicity, bilateral renal vascular disease, or systemic diseases (hepatorenal syndrome, glomerulonephritis, renal vasculitis, etc.)

--Prior/Concurrent Therapy--

Group 1: No recent immunosuppressive therapy Group 2 and 3: No prior renal transplantation No prior alpha-MSH Group 3: No prior dialysis for this episode of ARF No anticipated need for dialysis for at least 24 hours At least 12 hours since prior diuretics, mannitol, or dopamine At least 14 days since prior immunosuppressive drugs

--Patient Characteristics--

No recent infection No known reaction to Terumo T175 dialyzer Not a prisoner Not pregnant or nursing No allergy to drugs used in study Not mentally impaired Group 3: No severe nonrenal medical condition that would interfere with the study (e.g., terminal cancer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 1999-02; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Robert Toto, Study Chair — University of Texas
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas